CLINICAL TRIAL: NCT01837355
Title: Modulation of Intestinal and Pulmonary Inflammation by Lactobacillus Rhamnosus Diet Supplementation in Pediatric Cystic Fibrosis (MoHuM-1)
Brief Title: Modulation of Intestinal and Pulmonary Inflammation by Lactobacillus Diet Supplementation in Pediatric Cystic Fibrosis
Acronym: MoHuM-1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Collaborators: Swiss Federal Institute of Technology (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Christian R Kahlert, MD, Consultant Pediatric Infectious Diseases, Cantonal Hospital of St. Gallen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EKSG 12/129/1B
Record Dates: First submitted 2013-04-10; First posted 2013-04-23 (Estimated); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Inflammation; Cystic Fibrosis; Microbiota
MeSH Terms: conditions — Pneumonia; Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): placebo once daily for 12 weeks
  Interventions: Dietary Supplement: Placebo
- Lactobacillus rhamnosus (Experimental): lactobacillus rhamnosus once daily for 12 weeks
  Interventions: Dietary Supplement: Lactobacillus rhamnosus

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus
  Arms: Lactobacillus rhamnosus
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Pulmonary inflammation is an independent risk factor for disease progression in cystic fibrosis patients (CF). Yet, no effective treatment is known to reduce this detrimental inflammation. Dysbiosis of the gut microbiota has been linked to inflammation in several inflammatory diseases. As children with CF have different faecal microbiota from their healthy siblings, modulating gut microbiota by lactobacillus rhamnosus diet supplementation might be a strategy to target the inflammatory state in CF. Study subjects (CF or healthy control) will receive either placebo or lactobacillus rhamnosus once daily as dietary supplementation for 12 weeks. After a one-week washout phase, they will be switched for another 12 weeks to the other trial arm. Effect on in intestinal and pulmonary inflammation as well as clinical outcome will be studied.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe CF disease

Exclusion Criteria:

* acute gastroenteritis 2 weeks prior to inclusion
* chronic disease other than CF (except CF associated disorders)
* oral or parenteral antibiotics 2 weeks prior to inclusion
* systemic steroids 4 weeks prior to inclusion
* any probiotic intake

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2013-02-22 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline at w12 and w24 in fecal calprotectin levels | Baseline, week 12, week 24
  Baseline, week 12 change from baseline, week 24 change from week 12
Change from baseline at w12 and w24 in pulmonary calprotectin levels | Baseline, w12, w24
  Baseline, week 12 change from baseline, week 24 change from week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens's Hospital of Eastern Switzerland, Sankt Gallen, Canton of St. Gallen, Switzerland